CLINICAL TRIAL: NCT02295865
Title: A Phase 2 Multicenter, Randomized, Double-blind, Placebo-Controlled, Trial to Evaluate Toreforant (JNJ-38518168) for the Treatment of Subjects With Moderate to Severe Plaque-type Psoriasis
Brief Title: A Study to Evaluate Safety and Efficacy of Toreforant (JNJ-38518168) in Participants With Moderate to Severe Plaque-type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR106239; 38518168PSO2001 (Other: Janssen Research & Development, LLC); 2015-000277-12 (EudraCT Number)
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Psoriasis
Keywords: Psoriasis; Toreforant; JNJ-38518168
MeSH Terms: conditions — Psoriasis | interventions — toreforant

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (4):
- JNJ-38518168 60 mg (Experimental): Participants will receive two tablets of JNJ-38518168, 30 milligram (mg) each for a total of 60 mg, together with one 30 mg matching placebo tablet and one 3 mg matching placebo tablet, orally, once daily, for 12 Weeks.
  Interventions: Drug: JNJ-38518168 60 mg; Drug: Placebo
- JNJ-38518168 30 mg (Experimental): Participants will receive one tablet of JNJ-38518168, 30 mg, together with two 30 mg matching placebo tablets and one 3 mg matching placebo tablet, orally, once daily, for 12 Weeks.
  Interventions: Drug: JNJ-38518168 30 mg; Drug: Placebo
- JNJ-38518168 3 mg (Experimental): Participants will receive one tablet of JNJ-38518168, 3 mg, together with three 30 mg matching placebo tablets, orally, once daily, for 12 Weeks.
  Interventions: Drug: JNJ-38518168 3 mg; Drug: Placebo
- Placebo (Experimental): Participants will receive three tablets of JNJ-38518168, 30 mg matching placebo, together with one 3 mg matching placebo tablet, orally, once daily, for 12 Weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-38518168 60 mg — Two tablets of JNJ-38518168, 30 milligram (mg) each for a total of 60 mg, orally, once daily.
  Other Names: Toreforant
  Arms: JNJ-38518168 60 mg
Drug: JNJ-38518168 30 mg — One tablet of JNJ-38518168, 30 mg, orally, once daily.
  Other Names: Toreforant
  Arms: JNJ-38518168 30 mg
Drug: JNJ-38518168 3 mg — One tablet of JNJ-38518168, 3 mg, orally, once daily.
  Other Names: Toreforant
  Arms: JNJ-38518168 3 mg
Drug: Placebo — Matching Placebo either 30 mg tablet or 3 mg tablet will be administered orally.

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of JNJ-38518168 in participants with moderate to severe plaque-type psoriasis (common genetically determined, chronic, inflammatory skin disease characterized by rounded erythematous, dry, scaling patches).

DETAILED DESCRIPTION:
This is a randomized (study medication assigned to participants by chance), double-blind (neither the researchers nor the participants know what treatment the participant is receiving), parallel-group, placebo-controlled (an inactive substance; a pretend treatment [with no drug in it] that is compared in a clinical trial with a drug to test if the drug has a real effect) study. The study consists of Screening Phase (maximum of 42 days prior to Week 0), Treatment Phase (Week 0-12) and Follow-up Phase (up to Week 16). Participants will be randomly assigned to receive JNJ-38518168 (3 milligram [mg] or 30 mg or 60 mg) or placebo once daily. The initial group of the participants will be randomized to either JNJ-38518168 30 mg or placebo. The dose assignments for the subsequent participants will depend on the results of up to 2 interim analyses. Efficacy will be primarily assessed by percentage of participants who achieve a Psoriasis Area and Severity Index (PASI) 75 response at Week 12. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a diagnosis of plaque-type psoriasis (with or without psoriatic arthritis [PsA]) for at least 6 months before the first administration of study drug
* Participant must have a Psoriasis Area and Severity Index (PASI) Greater Than or equal to (>=) 12 at screening and at baseline
* Participant must have an Investigator's Global Assessment (IGA) >=3 at screening and at baseline
* A woman of childbearing potential must have a negative urine pregnancy test at screening and at Week 0
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control during the study and for 4 months after receiving the last administration of study drug. All men must also agree to not donate sperm during the study and for 4 months after receiving the last administration of study drug

Exclusion Criteria:

* Participant has a history or current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, cerebral, or psychiatric disease
* Participant has a current malignancy or history of malignancy within 5 years before screening (with the exception of a nonmelanoma skin cancer that has been adequately treated with no evidence of recurrence for at least 3 months before the first study drug administration, or cervical carcinoma in situ that has been treated with no evidence of recurrence for at least 1 year before the first study drug administration)
* Participant has a history of lymphoproliferative disease, including lymphoma; a history of monoclonal gammopathy of undetermined significance (MGUS); or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy or splenomegaly
* Participant has a history of chronic or recurrent infectious disease, including but not limited to chronic renal infection, chronic chest infection (eg, bronchiectasis), recurrent urinary tract infection (recurrent pyelonephritis or chronic nonremitting cystitis), fungal infection (mucocutaneous candidiasis), or open, draining, or infected skin wounds or ulcers
* Participant has a history of an infected joint prosthesis, or has received antibiotics for a suspected infection of a joint prosthesis, if that prosthesis has not been removed or replaced
* Participant has ever received any previous biologic therapy for psoriasis or psoriatic arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-11-17 (Actual); Primary Completion 2016-03-11 (Actual); Study Completion 2016-03-11 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve Psoriasis Area and Severity Index (PASI) 75 Response at Week 12 | Week 12
  The PASI score is a combined assessment of lesion severity and area affected into single score. Body will be divided into 4 sections:head, arms, trunk, and legs. For each section, percent (%) area of skin involved was estimated:0=0%, 1=less than (<) 10%, 2=10 to <30%, 3=30 to <50%, 4=50 to <70%, 5=70 to <90%, 6=90 to 100%. Severity will be estimated by clinical signs:erythema,induration,desquamation;scale:0= none to 4=maximum. Final PASI=sum of severity parameters for each section*area score*weight of section (head:0.1,arms:0.2,body:0.3,legs:0.4);total possible score range: 0=no disease to 72=maximal disease. A PASI 75 response defined as greater than or equal to (>=) 75 % improvement in PASI score from baseline.

SECONDARY OUTCOMES:
Percentage of Participants Who Achieve a Score of 0 or 1 on the Investigator's Global Assessment (IGA) at Week 12 | Week 12
  The IGA documents the investigator's assessment of the participants psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling on a scale of 0 to 4 (higher score = more severe). The participant's psoriasis is assessed as 5-point scale as follows: 0=cleared, 1=minimal, 2=mild, 3=moderate, 4=severe.
Percentage of Participants Who Achieve PASI 50, PASI 75, PASI 90 and PASI 100 Responses | Week 0, 2, 4, 6, 8, 12 and 16
  The PASI score is a combined assessment of lesion severity and area affected into single score. Body will be divided into 4 sections:head, arms, trunk, and legs. For each section, % area of skin involved was estimated:0=0%, 1= <10%, 2=10 to <30%, 3=30 to <50%, 4=50 to <70%, 5=70 to <90%, 6=90 to 100%. Severity will be estimated by clinical signs:erythema,induration,desquamation;scale:0= none to 4=maximum. Final PASI=sum of severity parameters for each section*area score*weight of section (head:0.1,arms:0.2,body:0.3,legs:0.4);total possible score range: 0=no disease to 72=maximal disease. A PASI 50, 75, 90, 100 response is defined as corresponding >= 50%, >=75%, >=90%, >=100% improvement in PASI score from baseline.
Percent Improvement From Baseline in PASI Score | Week 0 (Baseline), 2, 4, 6, 8, 12 and 16
  The PASI score is a combined assessment of lesion severity and area affected into single score. Body will be divided into 4 sections:head, arms, trunk, and legs. For each section, % area of skin involved was estimated:0=0%, 1= <10%, 2=10 to <30%, 3=30 to <50%, 4=50 to <70%, 5=70 to <90%, 6=90 to 100%. Severity will be estimated by clinical signs:erythema,induration,desquamation;scale:0= none to 4=maximum. Final PASI=sum of severity parameters for each section*area score*weight of section (head:0.1,arms:0.2,body:0.3,legs:0.4);total possible score range: 0=no disease to 72=maximal disease.
Percentage of Participants Who Achieve Investigator's Global Assessment (IGA) Score Responses of 0, 1 or 2; 0 or 1; and 0 | Week 0, 2, 4, 6, 8, 12 and 16
  The IGA documents the investigator's assessment of the participants psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling on a scale of 0 to 4 (higher score = more severe). The participant's psoriasis is assessed as 5-point scale as follows: 0=cleared, 1=minimal, 2=mild, 3=moderate, 4=severe.
Change From Baseline in Psoriasis Symptom and Sign Diary (PSSD) Symptom and Sign Score at Week 12 | Baseline and Week 12
  The PSSD is a questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered patient-reported outcome (PRO) instrument that includes 11 items covering symptoms and patient-observable signs. The psoriasis symptom score includes itch (Q1), pain (Q11), stinging (Q10), burning (Q9) and skin tightness (Q4) and average value of all 5 items will be converted into 0-100 score, where 0= least severe to 100=most severe. The psoriasis sign score includes skin dryness (Q2), cracking (Q3), scaling (Q5), shedding or flaking (Q6), redness (Q7) and bleeding (Q8) and average value of all 6 items will be converted into 0-100 score, where 0= least severe to 100=most severe. Total score includes all 11 individual items (both symptom and signs) and average value of all 11 items will be converted into 0-100 score, where 0= least severe to 100=most severe.
Percentage of Participants Who Achieve a PSSD Symptom Score of 0 or PSSD Sign Score of 0 at Week 12 | Week 12
  The PSSD is a questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms and patient-observable signs. The psoriasis symptom score includes itch (Q1), pain (Q11), stinging (Q10), burning (Q9) and skin tightness (Q4) and average value of all 5 items will be converted into 0-100 score, where 0= least severe to 100=most severe. The psoriasis sign score includes skin dryness (Q2), cracking (Q3), scaling (Q5), shedding or flaking (Q6), redness (Q7) and bleeding (Q8) and average value of all 6 items will be converted into 0-100 score, where 0= least severe to 100=most severe. Total score includes all 11 individual items (both symptom and signs) and average value of all 11 items will be converted into 0-100 score, where 0= least severe to 100=most severe.
Percentage of Participants who Achieve PSSD Individual (Psoriasis Symptom Score and Psoriasis Sign Score) Sub-Scale Score of 0 at Week 12 | Week 12
  The PSSD is a questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms and patient-observable signs. The psoriasis symptom score includes itch (Q1), pain (Q11), stinging (Q10), burning (Q9) and skin tightness (Q4) and average value of all 5 items will be converted into 0-100 score, where 0= least severe to 100=most severe. The psoriasis sign score includes skin dryness (Q2), cracking (Q3), scaling (Q5), shedding or flaking (Q6), redness (Q7) and bleeding (Q8) and average value of all 6 items will be converted into 0-100 score, where 0= least severe to 100=most severe. Total score includes all 11 individual items (both symptom and signs) and average value of all 11 items will be converted into 0-100 score, where 0= least severe to 100=most severe.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (13):
- United States (10):
  - Los Angeles, California
  - Santa Monica, California
  - Atlanta, Georgia
  - Indianapolis, Indiana
  - Plainfield, Indiana
  - Louisville, Kentucky
  - Portland, Oregon
  - Johnston, Rhode Island
  - San Antonio, Texas
  - Spokane, Washington
- Poland (3):
  - Bydgoszcz
  - Lodz
  - Warsaw